CLINICAL TRIAL: NCT00160758
Title: Physical Characteristics of Retrieved Massive Allografts
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 214-1999
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Bone Cancer
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: retrieve massive allograft — Allograft constructs removed because of infection or cancer complications will be retained for biomechanical testing

SUMMARY:
This purpose of this study is to measure the strength of tissue allografts that have been in the body various lengths of time.

DETAILED DESCRIPTION:
Allograft bone is the primary source of graft material for large skeletal defects resulting from trauma, disease, oncological resection, or reconstruction of failed total joint arthroplasties. The physical characteristics of such grafts after various intervals of remodeling and incorporation in vivo have never been studied.

The purpose of this study is to obtain tissue from allografts retrieved at autopsy, at amputation for oncological complications and from patients undergoing revision procedures for failed allograft transplantation. We will evaluate the mechanical properties, histomorphometric indices and presence of microfractures.

Our hypotheses are:

* histomorphometric parameters of porosity and microfracture density will predict allograft strength,
* microfracture density will be correlated with time in vivo and allograft strength,
* the rate of host-allograft nonunion and fracture will correlate with radiation therapy and chemotherapy.

The retrieved tissue will be processed using standard undecalcified histology and quantitatively assessed for degree of incorporation, allograft porosity, and microfracture density. The biomechanical characteristics of the bulk allograft and allograft-host junction will be quantified and compared to allograft bone prior to transplantation.

ELIGIBILITY:
Inclusion Criteria:

* failed allograft bone
* removal of allograft due to oncological complications
* amputation due to oncological complications

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Orthopaedic clinic
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 1999-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark T. Scarborough, M.D., Principal Investigator — University of Florida
Locations (1):
- UF Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States